CLINICAL TRIAL: NCT05734404
Title: Longitudinal Study for Central Nervous System Vasculitis
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: VCRC5509
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Central Nervous System Vasculitis; CNS Vasculitis; CNSV; Vasculitis
MeSH Terms: conditions — Vasculitis, Central Nervous System; Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary central nervous system vasculitis (CNSV) is a potentially fatal, single-organ vasculitis that often involves a spectrum of neurologic complications, including strokes, cognitive and speech impairment, visual loss, dementia, and encephalopathy. The purpose of this study is to establish a research cohort to investigate the disease process, treatments, and patient outcomes in CNSV.

DETAILED DESCRIPTION:
Primary central nervous system vasculitis (CNSV) is a potentially fatal, single-organ vasculitis that often involves a spectrum of neurologic complications, including strokes, cognitive and speech impairment, visual loss, dementia, and encephalopathy. Originally described in the early 1950s, research in the disease has been slow to progress, largely limited by the rarity of the disease and the lack of biologic materials for basic and translational investigations. To date, the bulk of research in the field has been clinical, largely consisting of retrospective case series, predominately from single sites, focusing on correlations among clinical, imaging, and histopathology data. Collectively these series suggest the existence of clinically-relevant subsets. Such studies, while enhancing our knowledge of this rare disease, are limited by small numbers of patients (especially those confirmed by histopathology), and the near absence of detailed investigations into the biomolecular and immunopathogenic basis of the disease.

Development of this longitudinal cohort and multicenter approach offers the potential to generate new insights, generate new questions, and further our understanding of its natural history, pathophysiology, genetic basis, and discovery of biomarkers to assess disease activity and prognosis.

Study visits will occur every 3 months for this first year, and then annually for two more years. Blood collection will occur at every visit. A physical exam and medical and medication history will at every visit; also, participants will be asked to complete several questionnaires to assess disease activity, health status, and tobacco, alcohol, and drug use.

ELIGIBILITY:
Inclusion Criteria:

i. Diagnostic criteria for CNSV

1. The presence of an acquired and otherwise unexplained neurologic deficit
2. The presence of either classic angiographic or histopathologic features of angiitis in the CNS
3. No evidence of systemic vasculitis or any condition that could cause the angiographic or pathologic features

ii. ≥18 years of age

Exclusion Criteria:

i. Unwilling to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with central nervous system vasculitis (CNSV). Enrollment will be sequential and participants will have disease in various stages and of different duration.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the pathogenesis of central nervous system vasculitis using disease history. | Study completion; from baseline through month 36.
  To study the manner of development of disease in patients affected with central nervous system vasculitis.

SECONDARY OUTCOMES:
PROMIS Questionnaires | Baseline, month 3, month 6, month 9, month 12, month 18, month 24, month 30, month 36
  Questions will ask about Cognition function on the PROMIS short form.
PROMIS Questionnaires | Baseline, month 3, month 6, month 9, month 12, month 18, month 24, month 30, month 36
  Questions will ask about depression on the PROMIS short form.
PROMIS Questionnaires | Baseline, month 3, month 6, month 9, month 12, month 18, month 24, month 30, month 36
  Questions will ask about fatigue on the PROMIS short form.
PROMIS Questionnaires | Baseline, month 3, month 6, month 9, month 12, month 18, month 24, month 30, month 36
  Questions will ask about Ability to participate in social roles and activities on the PROMIS short form.
PROMIS Questionnaires | Baseline, month 3, month 6, month 9, month 12, month 18, month 24, month 30, month 36
  Questions will ask about Upper extremity function on the PROMIS short form.
PROMIS Questionnaires | Baseline, month 3, month 6, month 9, month 12, month 18, month 24, month 30, month 36
  Questions will ask about lower extremity function on the PROMIS short form.
PROMIS Questionnaires | Baseline, month 3, month 6, month 9, month 12, month 18, month 24, month 30, month 36
  Questions will ask about Global Health (physical) on the PROMIS short form.
PROMIS Questionnaires | Baseline, month 3, month 6, month 9, month 12, month 18, month 24, month 30, month 36
  Questions will ask about Global Health (mental) on the PROMIS short form.

CONTACTS AND LOCATIONS:
Overall Officials: Rula Hajj-Ali, MD, Principal Investigator — The Cleveland Clinic; Leonard Calabrese, MD, Principal Investigator — The Cleveland Clinic; Peter Merkel, MD, Principal Investigator — University of Pennsylvania
Locations (6):
- United States (4):
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
- Canada (2):
  - St. Joseph's Healthcare, Hamilton
  - University of Toronto/Sinai Health, Toronto

IPD SHARING:
Plan to Share IPD: No